CLINICAL TRIAL: NCT05560815
Title: EPeCS - Epidemiology of Perioperative Care in Sweden 2015-2020
Brief Title: Epidemiology of Perioperative Care in Sweden
Acronym: EPeCS
Status: Active, not recruiting | Type: Observational
Sponsor: Linkoeping University (Other Government)
Collaborators: Region Östergötland (Other)
Responsible Party: Principal Investigator, Rasmus Åhman, Principal Investigator, Linkoeping University
Other Study IDs: EPeCS - ANOPIVA
Record Dates: First submitted 2022-09-22; First posted 2022-09-29 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Surgery
Keywords: Epidemiological study; Adverse effects; Operative surgical procedures; Perioperative process; Risk factors; Mortality; Postoperative complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- The Swedish surgical population: All adult patients (≥18 years) undergoing any surgical procedure registered in SPOR during 1 January 2015 - 31 December 2020.
  Interventions: Procedure: Any surgical procedure

INTERVENTIONS:
Procedure: Any surgical procedure — Might differ for substudies.

SUMMARY:
The Epidemiology of Perioperative Care in Sweden (EPeCS) study is a registry-based, retrospective extensive analysis of the whole adult (≥18 years) surgical population in Sweden during six full years, 1 January 2015 - 31 December 2020. Patients are retrieved from the Swedish Perioperative Registry (SPOR) which has full national coverage of public healthcare.

The study aspire to integrate pre-, peri- and postoperative components of the whole perioperative process as well as process, patient, anaesthesia and surgical factors. This allows for careful risk-adjustment and is a major strength of the project. This will require cross-matching data from several national quality registries.

EPeCS will serve as a database to be used as the foundation for several substudies that are to be conducted (10 at the present moment). Specific study focuses and aims are described in the "Detailed Description" section below.

The present study aims to provide a comprehensive audit of the surgical population in Sweden, and to identify factors that are of importance for outcome. The investigators aim to identify factors that will allow a better prediction of outcome, if they are modifiable, and if they are different for different lengths of follow-up. The ultimate goal is to provide hypotheses for directed therapies (eg. different types of anaesthesia), processes (eg. designated around-the-clock hip-fracture surgical teams), postoperative care (eg. extended PACU care instead of intensive care) in order to decrease suffering and increase cost-efficacy in Swedish healthcare.

DETAILED DESCRIPTION:
Specific aim for each substudy:

1. Epidemiology of Perioperative Care in Sweden
2. Risk factors for mortality after acute hip fracture surgery
3. Healthcare need after surgery
4. outcomes after urgent and emergency surgery
5. impact of estimated glomerular filtration rate (eGFR) on survival after elective surgery
6. effect of angiotensin receptor blocker (ARB) and angiotensin converting enzyme inhibitor (ACEi) non-resumption on postoperative outcome
7. impact of socioeconomic status
8. impact of university hospital status
9. effect of body mass index (BMI)
10. effect of post-anaesthesia care unit (PACU) stay

All these 10 specific areas have knowledge gaps regarding perioperative care.

Although there are 10 specific aims in this project, the same dataset (or parts thereof) from SPOR will be used for all substudies. The investigators will include all adult patients (≥18 years) undergoing any surgical procedure, except for the substudies where specific populations are prespecified, which are substudy 2: hip fracture surgery; substudy 4: urgent and emergency procedures; substudies 5,6 and 10: elective procedures with planned overnight stay; substudies 7 and 8: large joint surgery (hip and knee replacements), acute hip fracture surgery, colectomy, mastectomy, transurethral resection of the prostate (TUR-P) and prostatectomy.

Outcome measures might also differ between substudies.

National Quality Registries that will provide data for EPeCS, presented as "register (registry holder)":

* Swedish Perioperative Registry, SPOR (Uppsala Clinical Research Centre, UCR)
* Longitudinal integrated database for health insurance and labour market studies, LISA (Statistics Sweden)
* Swedish National Inpatient Register (the National Board of Health and Welfare)
* Swedish National Outpatient Register (the National Board of Health and Welfare)
* Swedish Drug Register (the National Board of Health and Welfare)
* Swedish Cause of death Register (the National Board of Health and Welfare)

The impetus for this project comes from the realization that surgery is not just a discrete event - it is part of a continuum of a larger journey of illness and health. The investigators hope to gain a comprehensive understanding of those patients who are at risk of poor outcome, their risk of death and burden of healthcare need after surgery.

Additional substudies might emerge.

ELIGIBILITY:
Inclusion Criteria:

* Underwent any surgical procedure in Sweden during the time period 1 Jan 2015 - 31 Dec 2020
* Registered in the Swedish Perioperative Registry (SPOR)
* ≥18 years of age
* Swedish social security number (to enable follow-up)

Exclusion Criteria:

* incorrect social security number
* incomplete mortality data
* the patient has chosen to opt-out of the register

The first two exclusion criteria are applied because they prevent correct follow-up of the primary outcome measure (mortality)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult (≥18 years) patients that have undergone any type of surgical procedure during 1 Jan 2015 - 31 Dec 2020 and are registered in the Swedish Perioperative Registry (SPOR).
Sampling Method: Probability Sample
Enrollment: 1500000 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
30-day mortality | Mortality up to 30 days post-surgery
  all cause
90-day mortality | Mortality up to 90 days post-surgery
  all cause
One-year mortality | Mortality up to one year post-surgery
  all cause
Two-year mortality | Mortality up to two years post-surgery
  all cause
Survival at longest follow-up | Longest possible follow-up post-surgery
  Survival rate through study completion, an average of 3 years

SECONDARY OUTCOMES:
Postoperative complications | 30 days (short-term) and one year (long-term) post-surgery, respectively
  Any new ICD10-SE code specified in SPOR
Healthcare need | Two years post-surgery
  Number of primary care visits
Critical Care need | 30 days post-surgery
  Admission to a critical care unit after surgery
Hospital readmission | 30 days post-surgery
  Readmission to hospital care after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Michelle S Chew, MD, PhD, Study Chair — Linkoeping University; Rasmus Åhman, MD, Principal Investigator — Linkoeping University
Locations (1):
- Department of Anaesthesia and Intensive Care, Linkoeping University Hospital, Linköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided